CLINICAL TRIAL: NCT01333033
Title: Randomized Phase II Trial of PET Scan-Directed Combined Modality Therapy in Esophageal Cancer
Brief Title: PET Scan Imaging in Assessing Response in Patients With Esophageal Cancer Receiving Combination Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80803; CDR0000698428 (Registry Identifier: NCI Physician Data Query); NCI-2011-02642 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer
Keywords: adenocarcinoma of the gastroesophageal junction; adenocarcinoma of the esophagus; stage IB esophageal cancer; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Carboplatin; Paclitaxel; Magnetic Resonance Spectroscopy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (FOLFOX regimen) (Experimental): Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin Calcium; Drug: Fluorouracil; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Radiation: Radiation Therapy
- Arm II (carboplatin + paclitaxel + radiation) (Experimental): Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Oxaliplatin — Given IV
  Arms: Arm I (FOLFOX regimen)
Drug: Leucovorin Calcium — Given IV
  Arms: Arm I (FOLFOX regimen)
Drug: Fluorouracil — Given IV
  Arms: Arm I (FOLFOX regimen)
Drug: Carboplatin — Given IV
Drug: Paclitaxel — Given IV
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Arms: Arm I (FOLFOX regimen)
Procedure: Computed Tomography — Undergo PET/CT scan
  Arms: Arm I (FOLFOX regimen)
Radiation: Radiation Therapy — Undergo RT

SUMMARY:
RATIONALE: PET scans done during chemotherapy may help doctors assess a patient's response to treatment and help plan the best treatment.

PURPOSE: This randomized phase II trial is studying PET scan imaging in assessing response in patients with esophageal cancer receiving combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To induce a complete pathologic response (pCR) rate of 20% in positron emission tomography (PET) scan non-responders treated with either induction FOLFOX or carboplatin/paclitaxel, who then crossover to the other regimen during radiotherapy.

Secondary

* To compare PET/CT response between induction treatment arms.
* To compare pCR between induction treatment arms among PET/CT scan responders.
* To directly compare pCR between induction treatment arms among non-responders if both treatment regimens are found to be efficacious.
* To determine 8-month progression-free survival (PFS) in PET/CT scan responders, and in non-responders treated with alternative crossover chemoradiotherapy.
* Estimate the PFS and overall survival (OS) curves, overall and among PET responders and PET/CT non-responders by induction treatment.
* To determine the rate of postoperative anastomotic leak after neoadjuvant chemotherapy followed by chemoradiation.
* To evaluate immunohistochemistry and RT-PCR of ERCC1, and genetic polymorphisms of ERCC1, XPD, and XRCC1.
* To evaluate status and levels of methylation of nine candidate biomarker genes as well as expression levels of selected specific microRNAs, which will be correlated with chemoradiation response.
* To compare the quality of life (QOL) of responders and nonresponders (as determined by PET/CT scanning) to presurgical treatment for esophageal cancer, in terms of global QOL, physical symptoms, physical functioning, and emotional well-being.
* To examine the association between OS and QOL in esophageal cancer patients treated with chemotherapy, chemoradiation therapy, and surgery.

OUTLINE: This is a multicenter study. Patients are stratified according to T-stage (T1-2 vs T3-4) and nodal status (N0 vs N+). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by ≥ 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent radiotherapy (RT) (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to arm II during RT.
* Arm II: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases ≥ 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to arm I during RT.

Within 4-10 weeks after completion of neoadjuvant chemoradiotherapy, patients undergo surgery at the discretion of the treating team.

Patients may undergo blood sample collection at baseline and periodically during study for correlative studies. Patients may also complete quality-of-life questionnaires at baseline and periodically during study.

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
* Surgically resectable, histologically confirmed esophageal adenocarcinoma, including Siewert gastroesophageal (GE) junction adenocarcinomas types 1 and 2
* T1N1-3M0 or T2-4NanyM0 as determined by endoscopic ultrasound (EUS) and PET/CT (histologic confirmation of lymph involvement is not required); all disease (tumor and nodes) must be both surgically resectable and capable of containment in a radiotherapy field; no T4 tumor with clear evidence of invasion of the vertebral column, heart, great vessels, or tracheobronchial tree
* All patients must have locoregional staging determined by endoscopic ultrasound (EUS) if technically feasible; endoscopy reports or subsequent gastrointestinal (GI) clinic note should clearly state both the T and N stage
* No evidence of distant metastases (as determined by EUS or PET/CT)
* Patients with cervical, supraclavicular, or other nodal disease that is either not included in the radiation field or is not able to be resected at the time of esophagectomy are not eligible
* Patient must have pre-resection tissue available for central pathology review, in case that the patient has a pCR at the time of surgical resection to confirm diagnosis
* Patients must have an fludeoxyglucose F 18 (FDG)-avid tumor with a maximum standard uptake value (SUVmax) of >= 5.0 on baseline PET/CT scan of primary tumor; baseline PET/CT scan should be performed; if it is necessary to repeat baseline PET/CT scan, reimbursement information is available
* No prior malignancy within 5 years of registration, with the exception of basal or squamous cell skin cancers, or in situ bladder or cervical cancer; patients with prior malignancy treated with surgery only and disease free for more than 5 years are eligible; however, no prior thoracic radiation therapy (RT) or abdominal RT or chemotherapy allowed
* No known contraindication to the use of fluorouracil, taxanes, or platinum compounds
* No history of severe hypersensitivity reaction to Cremophor EL
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must be non-pregnant and non-nursing; women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to randomization; women of child-bearing potential include any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >= 12 consecutive months; or women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35mIU/mL); even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential
* Absolute neutrophil count (ANC) >= 1,500/μL
* Platelet count >= 100,000/μL
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Calculated creatinine clearance >= 60 mL/min
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 times ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karyn A. Goodman, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (68):
- United States (68):
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin

REFERENCES:
- [Derived] Goodman KA, Ou FS, Hall NC, Bekaii-Saab T, Fruth B, Twohy E, Meyers MO, Boffa DJ, Mitchell K, Frankel WL, Niedzwiecki D, Noonan A, Janjigian YY, Thurmes PJ, Venook AP, Meyerhardt JA, O'Reilly EM, Ilson DH. Randomized Phase II Study of PET Response-Adapted Combined Modality Therapy for Esophageal Cancer: Mature Results of the CALGB 80803 (Alliance) Trial. J Clin Oncol. 2021 Sep 1;39(25):2803-2815. doi: 10.1200/JCO.20.03611. Epub 2021 Jun 2. PMID 34077237
- [Derived] Ku GY, Bains MS, Park DJ, Janjigian YY, Rusch VW, Rizk NP, Yoon SS, Millang B, Capanu M, Goodman KA, Ilson DH. Phase II study of bevacizumab and preoperative chemoradiation for esophageal adenocarcinoma. J Gastrointest Oncol. 2016 Dec;7(6):828-837. doi: 10.21037/jgo.2016.08.09. PMID 28078107

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOX Responder: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks.
- FOLFOX Non-Responder: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.n Emission Tomography: Undergo PET/CT scan
- CP Responder: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks.
- CP Non-Responder: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT
- CP No Cross-over: Carboplatin/ Paclitaxel days 1,8,22,29
- FOLFOX6 No Cross-over: modified FOLFOX6 days 1,15, 29
Period: Overall Study
Arm/Group | FOLFOX Responder | FOLFOX Non-Responder | CP Responder | CP Non-Responder | CP No Cross-over | FOLFOX6 No Cross-over
Started | 72 | 39 | 64 | 50 | 14 | 18
Completed | 72 | 39 | 64 | 50 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 14 | 18
Not completed — Ineligible | 0 | 0 | 0 | 0 | 6 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2
Not completed — PET inevaluable | 0 | 0 | 0 | 0 | 2 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Progression | 0 | 0 | 0 | 0 | 0 | 1
Not completed — MD Decision | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who enrolled on this trial are included in this analysis.
Groups:
- Arm I (FOLFOX Regimen): Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.
  Oxaliplatin: Given IV Leucovorin Calcium: Given IV Fluorouracil: Given IV Carboplatin: Given IV Paclitaxel: Given IV Positron Emission Tomography: Undergo PET/CT scan Computed Tomography: Undergo PET/CT scan Radiation Therapy: Undergo RT
- Arm II (Carboplatin + Paclitaxel + Radiation): Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT
  Carboplatin: Given IV Paclitaxel: Given IV Radiation Therapy: Undergo RT
- Total: Total of all reporting groups
Arm/Group | Arm I (FOLFOX Regimen) | Arm II (Carboplatin + Paclitaxel + Radiation) | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Continuous [Median (Full Range); unit: years] | 62 [22 to 84] | 64 [42 to 80] | 64 [22 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 113 | 114 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 126 | 124 | 250
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 4 | 10
  White | 119 | 116 | 235
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 129 | 128 | 257

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathological Response (pCR) of PET/CT Non-responders
Description: The primary endpoint of this study is the percentage of PET/CT non-responders within each induction treatment group reporting a pCR. A pCR is defined as having no tumor found on pathology review at surgery in all resected lymph nodes and tissue. All tissues sampled must have NO viable tumor.
Time Frame: Up to 5 years
Population: All eligible patients that registered to treatment and reported no PET/CT response to induction treatment were included in this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants with a pCR
Groups:
- FOLFOX Non-Responder: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.> >>>
  >
  >>> Oxaliplatin: Given IV>
  >>>
  >
  >>> Leucovorin Calcium: Given IV>
  >>>
  >
  >>> Fluorouracil: Given IV>
  >>>
  >
  >>> Carboplatin: Given IV>
  >>>
  >
  >>> Paclitaxel: Given IV>
  >>>
  >
  >>> Positron Emission Tomography: Undergo PET/CT scan>
  >>>
  >
  >>> Computed Tomography: Undergo PET/CT scan>
  >>>
  >
  >>> Radiation Therapy: Undergo RT
- CP Non-Responder: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT>
  >>>
  >
  >>> Carboplatin: Given IV>
  >>>
  >
  >>> Paclitaxel: Given IV>
  >>>
  >
  >>> Radiation Therapy: Undergo RT
Arm/Group | FOLFOX Non-Responder | CP Non-Responder
Number analyzed (Participants) | 39 | 50
percentage of participants with a pCR | 17.95 [7.54 to 33.53] | 20 [10.03 to 33.72]
Statistical Analysis 1: Comparison: FOLFOX Non-Responder vs CP Non-Responder; Test type: Superiority; p = 1.0, Fisher Exact

2. Secondary Outcome: PET/CT Response Between Treatment Arms
Description: A PET/CT response to induction therapy is defined as metabolic activity of the tumor decreasing by >=35%, as measured by maximum standardized uptake value (SUVmax).
Time Frame: Up to 5 years
Population: All participants that were assessed for an induction response are included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients with a response
Groups:
- FOLFOX Regimen: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.> >> >> >> > >> >> >> Oxaliplatin: Given IV> >> >> >> > >> >> >> Leucovorin Calcium: Given IV> >> >> >> > >> >> >> Fluorouracil: Given IV> >> >> >> > >> >> >> Carboplatin: Given IV> >> >> >> > >> >> >> Paclitaxel: Given IV> >> >> >> > >> >> >> Positron Emission Tomography: Undergo PET/CT scan> >> >> >>
  >
  >>
  >>
  >> Computed Tomography: Undergo PET/CT scan>
  >>
  >>
  >>
  >
  >>
  >>
  >> Radiation Therapy: Undergo RT
- CP (Carboplatin + Paclitaxel + Radiation): Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT>
  >>
  >>
  >>
  >
  >>
  >>
  >> Carboplatin: Given IV>
  >>
  >>
  >>
  >
  >>
  >>
  >> Paclitaxel: Given IV>
  >>
  >>
  >>
  >
  >>
  >>
  >> Radiation Therapy: Undergo RT
Arm/Group | FOLFOX Regimen | CP (Carboplatin + Paclitaxel + Radiation)
Number analyzed (Participants) | 111 | 114
percentage of patients with a response | 64.86 [55.23 to 73.69] | 56.14 [46.54 to 65.42]

3. Secondary Outcome: pCR Compared Between Induction Treatment Arms Among PET/CT Responders
Description: A PET/CT response to induction therapy is defined as metabolic activity of the tumor decreasing by >=35%, as>
  >>
  >>
  >> measured by maximum standardized uptake value (SUVmax). A pCR is defined as having no tumor found on pathology review at surgery in all resected lymph nodes and tissue. All tissues sampled must have NO viable tumor.
Time Frame: Up to 5 years
Population: All eligible patients that were assessed as a PET responder by induction were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants with a pCR
Groups:
- FOLFOX Responder: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.> >> >> >> > >> >> >> Oxaliplatin: Given IV> >> >> >> > >> >> >> Leucovorin Calcium: Given IV> >> >> >> > >> >> >> Fluorouracil: Given IV> >> >> >> > >> >> >> Carboplatin: Given IV> >> >> >> > >> >> >> Paclitaxel: Given IV> >> >> >> > >> >> >> Positron Emission Tomography: Undergo PET/CT scan> >> >> >>
  >
  >>
  >>
  >> Computed Tomography: Undergo PET/CT scan>
  >>
  >>
  >>
  >
  >>
  >>
  >> Radiation Therapy: Undergo RT
- CP (Carboplatin + Paclitaxel + Radiation) Responder: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT>
  >>
  >>
  >>
  >
  >>
  >>
  >> Carboplatin: Given IV>
  >>
  >>
  >>
  >
  >>
  >>
  >> Paclitaxel: Given IV>
  >>
  >>
  >>
  >
  >>
  >>
  >> Radiation Therapy: Undergo RT
Arm/Group | FOLFOX Responder | CP (Carboplatin + Paclitaxel + Radiation) Responder
Number analyzed (Participants) | 72 | 64
percentage of participants with a pCR | 40.28 [28.88 to 52.5] | 14.06 [6.64 to 25.02]

4. Secondary Outcome: pCR Compared Among Non-responders Between Induction Treatment Arms if Treatment Regimens Are Found to be Efficacious
Description: A Complete Pathological Response (pCR) is defined as having no tumor found on pathology review at surgery in all resected lymph nodes and tissue. All tissues sampled must have NO viable tumor. A non-responder was defined as having a PET/CT SUV (standard uptake value) decrease of less than 35% after induction.>
  >>>
  >
  >>> Among the patients who completed induction therapy and did not respond, the percentage of patients reporting a pCR in each arm were compared.
Time Frame: Up to 5 years
Population: All patients who completed induction therapy and were classified as a non-responder were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants with a pCR
Groups:
- FOLFOX Regimen Non-Responders: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.> >>>
  >
  >>> Oxaliplatin: Given IV>
  >>>
  >
  >>> Leucovorin Calcium: Given IV>
  >>>
  >
  >>> Fluorouracil: Given IV>
  >>>
  >
  >>> Carboplatin: Given IV>
  >>>
  >
  >>> Paclitaxel: Given IV>
  >>>
  >
  >>> Positron Emission Tomography: Undergo PET/CT scan>
  >>>
  >
  >>> Computed Tomography: Undergo PET/CT scan>
  >>>
  >
  >>> Radiation Therapy: Undergo RT
- CP (Carboplatin + Paclitaxel + Radiation) Non-Responders: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks. Patients without responsive disease (metabolic activity did not decrease by 35%) cross over to Arm I during RT>
  >>>
  >
  >>> Carboplatin: Given IV>
  >>>
  >
  >>> Paclitaxel: Given IV>
  >>>
  >
  >>> Radiation Therapy: Undergo RT
Arm/Group | FOLFOX Regimen Non-Responders | CP (Carboplatin + Paclitaxel + Radiation) Non-Responders
Number analyzed (Participants) | 39 | 50
percentage of participants with a pCR | 17.95 [7.54 to 33.53] | 20 [10.03 to 33.72]

5. Secondary Outcome: Progression Free Survival (PFS) Among PET/CT Non-responders Within Each Induction Treatment Group
Description: A non-responder was defined as having a PET/CT SUV (standard uptake value) decrease of less than 35% after induction.
  Among the patients who completed induction therapy and did not respond, the progression free survival in each arm were compared. PFS will be measured from study entry until documented progression or death from any cause. PFS will be estimated using the method of Kaplan and Meier.
Time Frame: Up to 5 years
Population: All patients that began induction therapy and did not report a response were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- FOLFOX Regimen Non-Responder: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreased by >= 35%) receive 3 additional courses of FOLFOX-6 therapy and undergo concurrent RT (3D-conformal or intensity-modulated) once daily, 5 days a week, for approximately 6 weeks. Patients without responsive disease (tumor metabolic activity did not decrease by 35%) cross over to Arm II during RT.
  >
  >>
  >
  >
  >>
  > Oxaliplatin: Given IV
  >
  >>
  >
  >
  >>
  > Leucovorin Calcium: Given IV
  >
  >>
  >
  >
  >>
  > Fluorouracil: Given IV
  >
  >>
  >
  >
  >>
  > Carboplatin: Given IV
  >
  >>
  >
  >
  >>
  > Paclitaxel: Given IV
  >
  >>
  >
  >
  >>
  > Positron Emission Tomography: Undergo PET/CT scan
  >
  >>
  >
  >
  >>
  > Computed Tomography: Undergo PET/CT scan
  >
  >>
  >
  >
  >>
  > Radiation Therapy: Undergo RT
Arm/Group | FOLFOX Regimen Non-Responder | CP Non-Responder
Number analyzed (Participants) | 39 | 50
months | NA [27.8 to NA] — Too few events have been recorded to estimate the median and upper confidence interval. | 33.4 [17.2 to NA] — Too few events have been recorded to estimate the upper confidence interval.

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- CP Non-Responder: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses. Patients then undergo PET/CT scan. Patients with responsive disease (tumor metabolic activity decreases >= 35%) continue to receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly for 5 weeks and undergo RT (3D-conformal or intensity-modulated) once a day, 5 days a week, for approximately 6 weeks.
- CP No Cross-over: Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 2 courses.
- FOLFOX No Cross-over: Patients receive modified FOLFOX-6 therapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 14 days for 3 courses.
Arm/Group | FOLFOX Responder | FOLFOX Non-Responder | CP Responder | CP Non-Responder | CP No Cross-over | FOLFOX No Cross-over
All-Cause Mortality (participants affected / at risk) | 3/72 | 1/39 | 2/64 | 4/49 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/72 | 1/39 | 2/64 | 4/49 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 72/72 | 38/39 | 63/64 | 46/49 | 9/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX Responder (N=72) | FOLFOX Non-Responder (N=39) | CP Responder (N=64) | CP Non-Responder (N=49) | CP No Cross-over (N=9) | FOLFOX No Cross-over (N=5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX Responder (N=72) | FOLFOX Non-Responder (N=39) | CP Responder (N=64) | CP Non-Responder (N=49) | CP No Cross-over (N=9) | FOLFOX No Cross-over (N=5)
Anemia (Blood and lymphatic system disorders) | 6 (19) | 7 (11) | 5 (9) | 10 (15) | 0 (0) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 (13) | 1 (5) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 4 (5) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (15) | 2 (2) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 36 (87) | 16 (24) | 23 (39) | 20 (42) | 1 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 10 (36) | 11 (28) | 7 (10) | 8 (19) | 1 (2) | 0 (0)
Esophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 6 (11) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jejunal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 56 (192) | 31 (88) | 42 (89) | 38 (120) | 6 (9) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 33 (66) | 18 (37) | 18 (29) | 20 (46) | 3 (5) | 1 (1)
Chills (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (39) | 9 (22) | 4 (4) | 6 (12) | 0 (0) | 0 (0)
Fever (General disorders) | 11 (16) | 4 (5) | 10 (15) | 8 (9) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 4 (14) | 4 (4) | 3 (5) | 2 (3) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (4) | 2 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 26 (66) | 15 (23) | 27 (37) | 19 (53) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 24 (46) | 18 (24) | 30 (50) | 15 (37) | 4 (4) | 0 (0)
Platelet count decreased (Investigations) | 44 (145) | 25 (52) | 44 (69) | 25 (71) | 2 (2) | 1 (1)
Weight loss (Investigations) | 4 (9) | 3 (3) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (4) | 8 (8) | 14 (16) | 1 (5) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (15) | 6 (7) | 2 (2) | 4 (5) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 5 (7) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (10) | 3 (3) | 4 (7) | 2 (11) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (7) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (16) | 3 (5) | 13 (25) | 5 (14) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (18) | 4 (7) | 11 (15) | 4 (6) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (27) | 6 (7) | 15 (26) | 3 (8) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 32 (120) | 16 (35) | 11 (30) | 12 (34) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 18 (37) | 5 (11) | 14 (21) | 4 (12) | 3 (7) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (36) | 10 (15) | 17 (30) | 21 (67) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 7 (26) | 4 (8) | 5 (8) | 5 (11) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (6) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (3) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less